CLINICAL TRIAL: NCT02886195
Title: EGFR-TKIs Combine Chemotherapy as First-line Therapy for Patients With Advanced EGFR Mutation-positive NSCLC
Acronym: effect
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: secgolc001
Record Dates: First submitted 2016-08-02; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-07

CONDITIONS: EGFR Gene Mutation
MeSH Terms: interventions — Pemetrexed; Cisplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PC plus erlotinib (Experimental): pemetrexed 500mg/m2 d1 plus cisplatin 80mg/m2 d1; concurrent erlotinib 150mg/d d1-21, per 3 week, for 4-6cycles, then erlotinib 150mg/d maintain therapy
  Interventions: Drug: pemetrexed; Drug: cisplatin; Drug: Erlotinib
- erlotinib (Active Comparator): erlotinib 150mg/d until "progress disease"
  Interventions: Drug: Erlotinib
- PC (Active Comparator): pemetrexed 500mg/m2 d1 plus cisplatin 80mg/m2 d1 for 4-6 cycles
  Interventions: Drug: pemetrexed; Drug: cisplatin

INTERVENTIONS:
Drug: pemetrexed — 500mg/m2 ivgtt d1, per three weeks
  Arms: PC; PC plus erlotinib
Drug: cisplatin — 80mg/m2 ivgtt d1, per three weeks
  Arms: PC; PC plus erlotinib
Drug: Erlotinib — 150mg po. every day
  Arms: PC plus erlotinib; erlotinib

SUMMARY:
The aim of this study was to compare the efficacy of EGFR-TKIs(Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitors) treatment plus concurrent chemotherapy versus sequential treatment with EGFR-TKIs and chemotherapy in patients with EGFR(Epidermal Growth Factor Receptor)-mutant non-small-cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is an open-label, randomized, parallel-group controlled clinical trial, and the study subjects recruited in this study are NSCLC patients mutant for EGFR gene (19del or L858R).

Subjects in the concurrent therapy group were given EGFR-TKIs treatment plus concurrent chemotherapy. Patients in the sequential treatment group were assigned to sequential EGFR-TKIs followed by chemotherapy group, which received TKIs monotherapy and then chemotherapy alone after disease progression; and sequential chemotherapy followed by EGFR-TKIs treatment, which was given first-line chemotherapy for 4 to 6 cycles, followed by maintenance therapy with EGFR-TKIs.

The endpoint of this study included clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Stage Ⅳ EGFR mutation-positive NSCLC
* Initial therapy
* ECOG performance status 0-1

Exclusion Criteria:

* EGFR mutation-negative
* Previous systemic antitumour treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months

SECONDARY OUTCOMES:
Response Rate (RR) | 2 months
Overall Survival (OS) | 6 months
Adverse Event (AE) | 2 months
  NCI CTC 4.03

CONTACTS AND LOCATIONS:
Overall Officials: zhiyong he he, master, Study Chair — Fujian province cancer hospital

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the process of the study

REFERENCES:
- [Derived] Lin J, Li M, Chen S, Weng L, He Z. Efficacy and Safety of First-Generation EGFR-TKIs Combined with Chemotherapy for Treatment-Naive Advanced Non-Small-Cell Lung Cancer Patients Harboring Sensitive EGFR Mutations: A Single-Center, Open-Label, Single-Arm, Phase II Clinical Trial. J Inflamm Res. 2021 Jun 16;14:2557-2567. doi: 10.2147/JIR.S313056. eCollection 2021. PMID 34168480